CLINICAL TRIAL: NCT00360763
Title: Study of Optimal Treatment Plan in Hypertensives With Anti-AT1-Receptor Autoantibody
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UH-01
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2006-08-07 (Estimated); Status verified 2006-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

INTERVENTIONS:
Drug: candesartan cilexetil

SUMMARY:
The autoantibodies against AT1 receptor (ATR-AA), behaving like an agonist were detected in patients with hypertension. ATR-AA which can blocked by ARB may play a role in the pathogenesis of hypertension. The present study is to explore whether AT1 receptor blocker has superior anti-hypertensive effect in patients with positive ATR-AA hypertension. Patients with 2 grade hypertension were recruited and ATR-AA was assayed by ELISA. A study was carried out and the efficacy of anti-hypertension was compared between candesartan cilexetil and ACE inhibitor imidapril.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension (2 grade)

Exclusion Criteria:

* Secondary hypertension
* Known sensitivity or intolerance to an angiotensin II receptor antagonist or ACE inhibitor
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hua Liao, Study Director — Union Hospital, Tongji Medical College
Locations (1):
- Department of Cardiology, Wuhan Union Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Liao YH, Wei YM, Wang M, Wang ZH, Yuan HT, Cheng LX. Autoantibodies against AT1-receptor and alpha1-adrenergic receptor in patients with hypertension. Hypertens Res. 2002 Jul;25(4):641-6. doi: 10.1291/hypres.25.641. PMID 12358154
- [Derived] Wei F, Jia XJ, Yu SQ, Gu Y, Wang L, Guo XM, Wang M, Zhu F, Cheng X, Wei YM, Zhou ZH, Fu M, Liao YH; SOT-AT1 Study Group. Candesartan versus imidapril in hypertension: a randomised study to assess effects of anti-AT1 receptor autoantibodies. Heart. 2011 Mar;97(6):479-84. doi: 10.1136/hrt.2009.192104. Epub 2011 Feb 4. PMID 21296780